CLINICAL TRIAL: NCT03068702
Title: New, Previously Unknown, Uses of Optical Coherence Tomography Angiography (OCTA): Sickle Cell Maculopathy
Brief Title: New, Previously Unknown, Uses of Optical Coherence Tomography Angiography (OCTA)
Acronym: OCTA
Status: Completed | Type: Observational
Sponsor: Dr. S.S. Michel Clinic (Other)
Responsible Party: Principal Investigator, Dr. Shawkat Michel, Principal Investigator, Dr. S.S. Michel Clinic
Other Study IDs: Optical Coherence Tomography
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Sickle Cell Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African Canadians: African Canadians with sickle cell disease maculopathy diagnosed by OCTA.
  Interventions: Device: Optical Coherence Tomography Angiography

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography

SUMMARY:
Sickle cell maculopathy was sparingly mentioned in the literature before despite the fact that sickle cell disease or sickle cell trait is common in people of many areas of the world. This study shows that OCTA is a very valuable, non invasive, office procedure that may well be used in diagnosing this disease.

DETAILED DESCRIPTION:
this is a clinical study of two African Canadian patients that were diagnosed with sickle cell trait. I used OCTA to show macular vascular occlusions that usually happen with this disease.

ELIGIBILITY:
Inclusion Criteria: people with sickle cell trait or sickle cell disease -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: African Canadian adults
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-08-21 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
vascular changes seen in the macular vasculature of people with sickle cell disease/ trait as compared to macular vasculature of normal macula. | through study completion, an average of one year
  in this angiography the delicate vasculature of the macula can be clearly visualized and documented.

CONTACTS AND LOCATIONS:
Overall Officials: shawkat s Michel, MD, FRCS Ed, Principal Investigator — Dr. S.S. Michel Clinic, 214 MHC, 156 street and 87 Ave, Edmonton, AB, Canada

IPD SHARING:
Plan to Share IPD: No